CLINICAL TRIAL: NCT03213431
Title: Assessing Patient-Reported Neurocognitive Functioning in Pediatric Oncology: A Pilot Study Toward Developing the Pediatric Neurocognitive Questionnaire (PNCQ)
Brief Title: Development of the Pediatric Neurocognitive Functioning Questionnaire
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PNCQ-HPP22
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Neurocognitive Disorders
Keywords: Cancer survivors; Instrument development; Neurocognitive functioning; Patient-reported outcomes; Qualitative interview
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IQ of <90 and ≥40: Patient-Reported Outcomes (PRO) will be evaluated in a group of 30 childhood cancer survivors with global neurocognitive impairment classified by IQ of <90 and ≥40 and 30 of their parents.
- IQ of ≥90: Patient-Reported Outcomes (PRO) will be evaluated in a group of 10 childhood cancer survivors with global neurocognitive unimpairment classified by IQ of ≥90 and 10 of their parents.

SUMMARY:
This study will examine self-reported neurocognitive functioning in pediatric cancer survivors whose cancer therapy may have included cranial radiation, intrathecal chemotherapy, and high-dose intravenous antimetabolite chemotherapy. There is evidence that these therapies which are directed at the central nervous system (CNS) can lead to reduced volumes of normal-appearing white matter and neurocognitive dysfunction.

Neurocognitive deficits can significantly impact pediatric cancer survivors' academic success, daily functional status, and quality of life. Previous studies demonstrate the need for screening and treating neurocognitive dysfunction in childhood cancer patients and survivors.

This pilot study will conduct cognitive debriefing tests with childhood cancer survivors, 30 with and 10 without neurocognitive deficits, and their parents. The collected data will aid in developing a comprehensive patient-reported outcomes (PRO) toolkit consisting of generic and specific cognitive and behavioral domains that are content-appropriate and interface-friendly for pediatric cancer populations.

PRIMARY OBJECTIVE:

* To conduct cognitive debriefing tests with 30 pediatric cancer survivors who have global neurocognitive impairment (i.e., the impaired group) to understand the cognitive process of answering the extant pediatric PRO measures by different levels of general intelligence quotient (IQ). Additionally, 10 pediatric cancer survivors who have at least average general IQ (i.e., the unimpaired group) will be recruited for a comparison purpose.

SECONDARY OBJECTIVE:

* To conduct semi-structured interviews with 30 parents/legal guardians of individuals who have global cognitive impairment as described in the primary objective in order to explore the general concept of their child's neurocognitive functioning, to rank the relative importance of different neurocognitive functioning domains, to inform a strategy for communicating with children and adolescents with impaired neurocognitive functioning for PRO research, and to suggest a user-friendly interface to collect PRO data from cognitively impaired children and adolescents. Additionally, 10 parents/legal guardians of individuals at least average general IQ will be recruited for comparison.

DETAILED DESCRIPTION:
Pediatric participants will undergo a 30-45 minute cognitive interview including three sections:

1. Introduction to the study and warm-up debriefing exercise.
2. Determination of participant's level of understanding by arranging circles of different sizes.
3. Completion of individual surveys including the Child Health & Illness Profile-Child Edition/Child Report Form (CHIP-CE/CRF), the Applied Cognition scale of the Neuro-QOL, and the Pediatric Perceived Cognitive Function (PedPCF - Child).

For patient participants who have not had IQ testing within the prior 3 years, IQ testing may be repeated.

Semi-structured interviews will be conducted with parents/legal guardians of pediatric participants including:

1. Open-ended questions to help researchers understand whether their child is able to complete the CHIP-CE/CRF, Applied Cognition scale of the Neuro-QOL, and the PedPCF - Child.
2. Concerns they may have about cognitive functioning issues and its importance for their child. They will also be asked their thoughts on how to communicate and interact effectively with children and adolescents who have cognitive delays and their feedback about a user-friendly way to collect patient-reported health data.
3. The pediatric participant responses will be compared with their parent/legal guardian responses to confirm the answers were accurate and to evaluate whether the child can recall appropriate information for a given time frame.

Interviews will be conducted primarily on the St. Jude campus, or via Skype video meeting as a secondary option.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivors who are off cancer therapies;
* Children/youth age 8-17.9 years and their parents/legal guardians (i.e. dyads);
* Impaired and unimpaired general IQs (IQ 40-89 for impaired and IQ ≥90 for unimpaired); AND
* English speaking participants.

Exclusion Criteria:

* Only the child/adolescent or the parent is able to participate (i.e. non-dyads);
* Severe/profound IQ deficits (IQ <40); AND
* Non-English speaking participants.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be childhood cancer survivors who are active After Completion of Therapy (ACT) patients consented to the SJLIFE clinical protocol and their parent/legal guardian.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Number of participants who are capable of completing the survey | At completion of the survey, up to 6 months after study enrollment.
  Capability will be defined as the number of participants who complete the survey based on comprehension for the content of survey items.

CONTACTS AND LOCATIONS:
Overall Officials: I-Chan Huang, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols